CLINICAL TRIAL: NCT00634751
Title: A Phase I/II STudy of Oxaliplatin, Oral Capecitabine and Sorafenib in Patients With Advanced Pancreatic and Biliary Carcinoma"
Brief Title: CO07204-Phase I/II of Oxaliplatin, Capecitabine & Sorafenib for Advanced Pancreatic & Biliary Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Bayer (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0248; CO07204 (Other: University of Wisconsin Carbone Cancer Center); H-2007-0248 (Other: Institutional Review Board); NCI-2011-00475 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Results first posted 2017-08-08 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2017-07

CONDITIONS: Pancreatic Neoplasms; Bile Duct Neoplasms
Keywords: advanced pancreatic and biliary tract carcinomas
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms | interventions — Oxaliplatin; Capecitabine; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I: 200mg Sorafenib+2DOC (Experimental): Cohort 1: 200mg Sorafenib+2DOC
  Oxaliplatin + Oral Capecitabine + Sorafenib
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Sorafenib
- Phase I: 400mg Sorafenib BID+2DOC (Experimental): Cohort 2: 400mg Sorafenib+2DOC
  Oxaliplatin + Oral Capecitabine + Sorafenib
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Sorafenib
- Phase II: Pancreatic Cancer (Experimental): Oxaliplatin + Oral Capecitabine + Sorafeni
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Sorafenib
- Phase II: Biliary Tract Cancer (Experimental): Oxaliplatin + Oral Capecitabine + Sorafeni
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Sorafenib

INTERVENTIONS:
Drug: Oxaliplatin — On days 1 and 15 of each 28 day treatment cycle, patients receive oxaliplatin 85 mg/m2 as a 2-hour IV infusion. Following the infusion of oxaliplatin, the infusion line should be flushed with Dextrose 5% in Water.
Drug: Capecitabine — Each course of oral capecitabine administration will commence following administration of oxaliplatin. Capecitabine 2250 mg/m2 will be given every 8 hours for a total of 6 doses as above, commencing with each cycle of therapy. Because capecitabine is provided in fixed dose forms, rounding will be necessary. Rounding will be to the nearest 150 mg on a per dose basis.
Drug: Sorafenib — Cohort 1 will receive 200 mg of sorafenib orally twice daily, cohort 2 will receive 400 mg orally twice daily, both beginning on the first day of the first cycle (see section 9.1). If needed, cohort -1 will be used, at 200 mg of sorafenib once daily. Sorafenib should be taken without food (at least 1 hour before or 2 hours after eating).
  Cohort I (Dose escalation phase) Agent Dose Route Day Cycle length
  Sorafenib 200 mg BID Oral Daily Every 28 days
  If 1/3 patients develop a DLT, enroll 3 patients at dose level -1 Sorafenib 200 mg po qd.
  Cohort II (Phase II studies at MTD) Agent Dose Route Day Cycle length
  Sorafenib 400 mg BID Oral Daily Every 28 days

SUMMARY:
This study involves the use of oxaliplatin, capecitabine, and sorafenib which are all drugs approved by the Food and Drug Administration (FDA) for use in the treatment of different cancers. Their use in this exact combination is considered experimental for the treatment of pancreas and biliary tract; however the combination has been tested in a preliminary trial. We are also testing a survey designed. The purpose of this research study is to investigate the chemotherapy drug sorafenib in combination with oxaliplatin and capecitabine chemotherapies for the treatment of pancreas and biliary tract cancers.to help patients report their side effects from chemotherapy treatments.

DETAILED DESCRIPTION:
Primary Objectives

* To assess the overall safety of sorafenib when administered with "the 2DOC regimen" capecitabine and oxaliplatin in patients with advanced or metastatic pancreas or biliary tract cancers.
* To define the dose limiting toxicity and maximally tolerated dose of this combination.
* To assess the clinical response rate (stable, partial and complete responses) of the combination in patients with advanced or metastatic pancreas or biliary tract cancers.

Secondary Objectives

* To define the time to progression and overall survival for patients treated with this regimen.
* To evaluate the congruency of the Adverse Events Self-Report Survey in determining patient reported side effects of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed locally advanced inoperable or metastatic adenocarcinoma of the pancreas or biliary tract who have not previously received more than one systemic treatment for their disease.
* Age at least 18 years old
* ECOG performance status 0-2.
* Patients must have adequate organ and marrow function as defined below:
* WBC at least 3,000
* ANC at least 1,500
* PLT at least 100,000
* total bilirubin must be less than 2.5 x institutional upper limit of norm
* AST(SGOT)/ALT(SGPT) must be less than 5 X institutional upper limit of normal
* creatinine clearance must be greater than 50 mL/min as calculated by the Cockroft-Gault formula
* Patients with ≤ grade 2 (CTC 3.0) neuropathy.
* At least one measurable lesion as defined by RECIST criteria
* The effects of oxaliplatin, capecitabine and sorafenib on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because DNA alkylating agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Because the risk of toxicity in nursing infants secondary to oxaliplatin treatment of the mother is unknown but may be harmful, breastfeeding should be discontinued if the mother is treated with oxaliplatin.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* No concomitant radiation therapy, or other systemic cancer therapies.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other toxicities.
* History of allergy to platinum compounds, capecitabine, sorafenib or to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, thrombolic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months, symptomatic congestive heart failure, unstable angina pectoris within 3 months prior to entry study, myocardial infarction within 6 months prior to study entry, ongoing cardiac arrhythmia (excluding atrial fibrillation), uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg, despite optimal medical management), pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug, or any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug, serious non-healing wound, ulcer, or bone fracture, evidence or history of bleeding diathesis or coagulopathy.
* Pregnant or nursing women are excluded from this study because oxaliplatin, capecitabine and sorafenib is a DNA alkylating agent with the potential for teratogenic or abortifacient effects. Female patients of reproductive potential must have a negative urine or serum pregnancy test within two weeks prior to enrolling.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Because of drug interactions with sorafenib, use of St. John's Wort or rifampin (rifampicin) is contraindicated. Patients may discontinue the use of these drugs to become eligible for the study
* Any condition that impairs patient's ability to swallow whole pills.
* HIV-positive patients receiving anti-retroviral therapy (HAART) are excluded from the study because of possible pharmacokinetic interactions.
* Second malignancy within the past 3 years (excluding nonmelanoma skin cancer and in situ cancers) that has not been treated with curative intent and is not currently without evidence of disease,
* Patients with known gastrointestinal malabsorption syndromes are excluded as this concurrent illness will affect absorption of the oral medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle K LoConte, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study accrued through the Wisconsin Oncology Network (WON), a network of academic and private practice institutions across the state of Wisconsin and the upper Midwest.
Groups:
- Phase I: 200mg Sorafenib+2DOC: Cohort 1: 200mg Sorafenib+2DOC
  Oxaliplatin + Oral Capecitabine + Sorafenib
  Oxaliplatin: Days 1 and 15 of each 28 day treatment cycle, patients receive oxaliplatin 85 mg/m2 as a 2-hour IV infusion. Next, the infusion line should be flushed with Dextrose 5% in Water.
  Capecitabine: Oral capecitabine administration will start after administration of oxaliplatin. Capecitabine 2250 mg/m2 will be given every 8 hours for a total of 6 doses, commencing with each cycle of therapy. Capecitabine is provided in fixed dose forms, and rounding will be to the nearest 150 mg on a per dose basis.
  Sorafenib: 200 mg of sorafenib orally twice daily, beginning on the first day of the first cycle. If needed, cohort -1 will be used, at 200 mg of sorafenib once daily.
  Cohort I
  Sorafenib 200 mg BID Oral Daily Every 28 days
  If 1/3 patients develop a DLT, enroll 3 patients at dose level -1 Sorafenib 200 mg po qd.
- Phase I: 400mg Sorafenib BID+2DOC: Cohort 2: 400mg Sorafenib+2DOC
  Oxaliplatin + Oral Capecitabine + Sorafenib
  Oxaliplatin: Days 1 and 15 of each 28 day treatment cycle, patients receive oxaliplatin 85 mg/m2 as a 2-hour IV infusion. Next, the infusion line should be flushed with Dextrose 5% in Water.
  Capecitabine: Oral capecitabine administration will start after administration of oxaliplatin. Capecitabine 2250 mg/m2 will be given every 8 hours for a total of 6 doses, commencing with each cycle of therapy. Capecitabine is provided in fixed dose forms, and rounding will be to the nearest 150 mg on a per dose basis.
  Sorafenib: 400 mg of sorafenib orally twice daily, both beginning on the first day of the first cycle (see section 9.1). If needed, cohort -1 will be used, at 200 mg of sorafenib once daily.
  Cohort II (Phase II studies at MTD) Agent Dose Route Day Cycle length
  Sorafenib 400 mg BID Oral Daily Every 28 days
- Phase II: Pancreatic Cancer; Phase II: Biliary Tract Cancer: Oxaliplatin + Oral Capecitabine + Sorafeni
  Oxaliplatin: Days 1 and 15 of each 28 day treatment cycle, patients receive oxaliplatin 85 mg/m2 as a 2-hour IV infusion. Next, the infusion line should be flushed with Dextrose 5% in Water.
  Capecitabine: Oral capecitabine administration will start after administration of oxaliplatin. Capecitabine 2250 mg/m2 will be given every 8 hours for a total of 6 doses, commencing with each cycle of therapy. Capecitabine is provided in fixed dose forms, and rounding will be to the nearest 150 mg on a per dose basis.
  Sorafenib: 400 mg of sorafenib orally twice daily, both beginning on the first day of the first cycle (see section 9.1). If needed, cohort -1 will be used, at 200 mg of sorafenib once daily.
Period: Phase I: 200mg Sorafenib+2DOC
Arm/Group | Phase I: 200mg Sorafenib+2DOC | Phase I: 400mg Sorafenib BID+2DOC | Phase II: Pancreatic Cancer | Phase II: Biliary Tract Cancer
Started | 9 | 0 | 0 | 0
Completed | 8 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Period: Phase I: 400mg Sorafenib BID+2DOC
Arm/Group | Phase I: 200mg Sorafenib+2DOC | Phase I: 400mg Sorafenib BID+2DOC | Phase II: Pancreatic Cancer | Phase II: Biliary Tract Cancer
Started | 0 | 7 | 0 | 0
Completed | 0 | 6 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Period: Pancreatic and Bilial Tract Cancer
Arm/Group | Phase I: 200mg Sorafenib+2DOC | Phase I: 400mg Sorafenib BID+2DOC | Phase II: Pancreatic Cancer | Phase II: Biliary Tract Cancer
Started | 0 | 0 | 24 | 8
Completed | 0 | 0 | 23 | 7
Not Completed | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants with histologically or cytologically confirmed adenocarcinoma of the pancreas or biliary tract were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: 200mg Sorafenib+2DOC | Phase I: 400mg Sorafenib BID+2DOC | Phase II: Pancreatic Cancer | Phase II: Biliary Tract Cancer | Total
Number analyzed (Participants) | 9 | 7 | 24 | 8 | 48
Age, Customized [Count of Participants; unit: Participants]
  =< 50 years of age | 1 | 1 | 1 | 2 | 5
  50-59 years of age | 1 | 2 | 8 | 2 | 13
  60-69 years of age | 3 | 4 | 7 | 2 | 16
  70-79 years of age | 3 | 0 | 7 | 2 | 12
  >= 80 years of age | 1 | 0 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 11 | 3 | 22
  Male | 4 | 4 | 13 | 5 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 7 | 21 | 5 | 41
  Unknown or Not Reported | 1 | 0 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 9 | 6 | 24 | 7 | 46
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 24 | 8 | 48

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Response rate of participant to treatment
Time Frame: Up to 18 months
Measure: Number; unit: participants
Groups:
- Phase II: Pancreatic Cancer; Phase II: Biliary Tract Cancer: Oxaliplatin + Oral Capecitabine + Sorafeni
  Oxaliplatin: Days 1 and 15 of each 28 day treatment cycle, patients receive oxaliplatin 85 mg/m2 as a 2-hour IV infusion. Next, the infusion line should be flushed with Dextrose 5% in Water.
  Capecitabine: Oral capecitabine administration will start after administration of oxaliplatin. Capecitabine 2250 mg/m2 will be given every 8 hours for a total of 6 doses, commencing with each cycle of therapy. Capecitabine is provided in fixed dose forms, and rounding will be to the nearest 150 mg on a per dose basis.
  Sorafenib: 200mg of sorafenib orally twice daily, both beginning on the first day of the first cycle.
Arm/Group | Phase I: 200mg Sorafenib+2DOC | Phase I: 400mg Sorafenib BID+2DOC | Phase II: Pancreatic Cancer | Phase II: Biliary Tract Cancer
Number analyzed (Participants) | 7 | 3 | 20 | 7
participants
  Partial Response | 1 | 1 | 3 | 1
  Stable Disease | 5 | 2 | 11 | 5
  Progressive Disease | 1 | 0 | 6 | 1

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Time to progression, defined as number of days from day of first study drug administration to the day the patient experiences an event of disease progression or death; summarized using point estimates of the median time to progression and associated 95% confidence intervals for each stratum separately.
Time Frame: Up to 18 months
Population: PFS was not a pre-specified Phase I outcome, and no data was collected or analyzed. No data was collected for Phase II biliary tract participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I: 200mg Sorafenib+2DOC | Phase I: 400mg Sorafenib BID+2DOC | Phase II: Pancreatic Cancer | Phase II: Biliary Tract Cancer
Number analyzed (Participants) | 0 | 0 | 19 | 0
Months |  |  | 6.0 [2.5 to 9.6] |

3. Secondary Outcome: Overall Survival
Description: Overall survival, defined as number of days from the day of first study drug administration to the day the patient dies, summarized using point estimates of the median time to progression, and associated 95% confidence intervals
Time Frame: Up to 18 months
Population: Overall survival was not a pre-specified Phase I outcome, and no data was collected or analyzed. No data was collected for Phase II biliary tract participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I: 200mg Sorafenib+2DOC | Phase I: 400mg Sorafenib BID+2DOC | Phase II: Pancreatic Cancer | Phase II: Biliary Tract Cancer
Number analyzed (Participants) | 0 | 0 | 19 | 0
Months |  |  | 8.1 [3.5 to 10.9] |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 years and 5 months.
Arm/Group | Phase I: 200mg Sorafenib+2DOC | Phase I: 400mg Sorafenib BID+2DOC | Phase II: Pancreatic Cancer | Phase II: Biliary Tract Cancer
Serious Adverse Events (participants affected / at risk) | 4/9 | 3/7 | 14/24 | 7/8
Other Adverse Events (participants affected / at risk) | 9/9 | 7/7 | 24/24 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: 200mg Sorafenib+2DOC (N=9) | Phase I: 400mg Sorafenib BID+2DOC (N=7) | Phase II: Pancreatic Cancer (N=24) | Phase II: Biliary Tract Cancer (N=8)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0
Allergic reaction/hypersensitivity (Immune system disorders) | 0 | 0 | 1 (1) | 0
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1) | 0 | 1 (1) | 0
Confusion (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Death (Gastrointestinal disorders) | 0 | 1 | 5 | 2
Dehydration (Gastrointestinal disorders) | 2 (2) | 0 | 0 | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Distension/bloating (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 — Abdominal
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Edema (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 | 0 — Limb
Fatigue (General disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 0 | 0 | 2 (2) | 0
Hemorrhage (Blood and lymphatic system disorders) | 0 | 0 | 2 (2) | 0
Hypotension (Cardiac disorders) | 1 (1) | 1 (1) | 0 | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 2 (2) | 0
Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
INR (International Normalized Ratio of Prothrombin Time) (Investigations) | 1 (1) | 0 | 1 (1) | 0
Intra-operative injury (Surgical and medical procedures) | 0 | 0 | 1 (1) | 0 — Duodenum
Liver dysfunction/failure (Hepatobiliary disorders) | 1 (1) | 0 | 0 | 0
Mucositis/stomatitis (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (3) | 0 | 0 | 1 (1)
Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 6 (6) | 0
Perforation (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1) — 1 duodenum; 1 gallbladder
Platelets (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1)
Rigors/chills (General disorders) | 0 | 0 | 1 (1) | 0
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Stricture/stenosis (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 — Duodenum
Syncope (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Thrombosis (Vascular disorders) | 1 (1) | 0 | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: 200mg Sorafenib+2DOC (N=9) | Phase I: 400mg Sorafenib BID+2DOC (N=7) | Phase II: Pancreatic Cancer (N=24) | Phase II: Biliary Tract Cancer (N=8)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 10 (23) | 5 (20)
Alkaline phosphatase (Investigations) | 5 (5) | 3 (3) | 11 (26) | 6 (18)
Allergic reaction (Immune system disorders) | 0 | 0 | 2 (2) | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (10) | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 (4) | 1 (2) | 8 (15) | 2 (3)
Amylase (Investigations) | 1 (1) | 0 | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 4 (7) | 0 | 11 (30) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 2 (3)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 | 0 | 11 (18) | 6 (18)
Ataxia (Nervous system disorders) | 0 | 0 | 1 (5) | 0
Auditory/ear - hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1 (1) | 0
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (2) | 1 (1) | 3 (3) | 4 (6)
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 2 (5) | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2) | 0 | 8 (12) | 3 (10)
Confusion (Psychiatric disorders) | 0 | 0 | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6) | 2 (3) | 8 (19) | 4 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 2 (2) | 0
CPK (creatine phosphokinase) (Investigations) | 1 (1) | 0 | 0 | 0
Creatinine (Investigations) | 2 (2) | 0 | 0 | 2 (7)
Dehydration (Metabolism and nutrition disorders) | 0 | 1 (1) | 3 (6) | 2 (2)
Dermal change lymphedema, phlebolymphedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0
Dermatology - peeling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 1 (2) | 0
Diarrhea (Gastrointestinal disorders) | 6 (15) | 5 (6) | 12 (27) | 3 (5)
Distension/bloating (Gastrointestinal disorders) | 0 | 0 | 1 (3) | 0
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 | 3 (3)
Dry eye syndrome (Eye disorders) | 0 | 0 | 1 (2) | 0
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (11) | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 4 (14) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 | 5 (10) | 1 (1)
Edema (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 4 (6) | 2 (4)
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 2 (2) | 0
Fatigue (General disorders) | 7 (19) | 4 (5) | 7 (9) | 8 (15)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 2 (2) | 2 (3)
Fistula, GI - Pancreas (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 (2) | 0
Flushing (Vascular disorders) | 0 | 0 | 1 (1) | 0
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 0 | 4 (12) | 0
Glomerular filtration rate (Renal and urinary disorders) | 0 | 0 | 0 | 1 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (5) | 1 (1) | 15 (53) | 6 (27)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 2 (11) | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 | 2 (3) | 0
Hemoglobin (Investigations) | 6 (10) | 4 (11) | 14 (33) | 4 (12)
Hemorrhage/bleeding (Blood and lymphatic system disorders) | 0 | 1 (1) | 2 (3) | 1 (5)
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Hot flashes/flushes (Vascular disorders) | 0 | 0 | 3 (5) | 0
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 2 (3) | 5 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1)
Hypotension (Vascular disorders) | 0 | 0 | 3 (4) | 0
Ileus, Ascites, Abdominal Pain, Anorexia, Oliguria (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Infection (Infections and infestations) | 3 (4) | 1 (1) | 4 (8) | 3 (5)
INR (Investigations) | 1 (1) | 1 (2) | 0 | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 | 1 (2)
Intra-operative injury - NERVES: CN V (trigeminal) sensory (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Jaundice (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1)
LDH (Investigations) | 0 | 0 | 1 (1) | 0
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (5) | 2 (2) | 10 (25) | 2 (22)
Lipase (Investigations) | 0 | 1 (1) | 4 (5) | 4 (8)
Liver dysfunction (Hepatobiliary disorders) | 1 (1) | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 5 (12) | 1 (8)
Magnesium, serum-low (Metabolism and nutrition disorders) | 0 | 0 | 3 (4) | 1 (1)
Mood alteration (Psychiatric disorders) | 1 (1) | 0 | 2 (5) | 0
Mucositis/stomatitis (Gastrointestinal disorders) | 2 (3) | 4 (5) | 5 (9) | 2 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 | 5 (13) | 2 (2)
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 (9) | 0
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (32) | 3 (4) | 10 (32) | 5 (8)
Neurology (Nervous system disorders) | 0 | 6 (6) | 2 (4) | 0
Neuropathy: sensory (Nervous system disorders) | 5 (10) | 0 | 14 (33) | 5 (17)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4 (4) | 0 | 6 (11) | 2 (19)
Obstruction, GI (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Ocular/visual - other (Eye disorders) | 0 | 0 | 1 (1) | 0
Pain (General disorders) | 9 (18) | 6 (11) | 17 (43) | 5 (12)
Palpitations (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Pancreatic endocrine: glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0
Perforation (Gastrointestinal disorders) | 0 | 0 | 1 (2) | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 2 (2) | 4 (6) | 2 (9)
Photosensitivity (Eye disorders) | 0 | 0 | 0 | 1 (1)
Platelets (Blood and lymphatic system disorders) | 5 (13) | 4 (11) | 15 (49) | 7 (29)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1)
Potassium, serum-low (hypokalemia) (Investigations) | 3 (5) | 3 (3) | 6 (17) | 2 (5)
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 5 (5) | 1 (4)
PTT (Investigations) | 0 | 0 | 1 (1) | 0
Rash (Skin and subcutaneous tissue disorders) | 2 (8) | 2 (2) | 5 (10) | 4 (13)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (3) | 8 (20) | 2 (8)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
Rigors/chills (General disorders) | 1 (1) | 0 | 3 (3) | 1 (1)
Seizure (Nervous system disorders) | 0 | 0 | 1 (2) | 0
Sinus drainage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (11) | 3 (11)
Stricture/stenosis (including anastomotic), GI - Biliary tree (Hepatobiliary disorders) | 1 (1) | 0 | 1 (1) | 0
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 (2)
Sweating (diaphoresis) (General disorders) | 3 (3) | 0 | 2 (4) | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Taste alteration (Gastrointestinal disorders) | 1 (2) | 0 | 4 (14) | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 0 | 3 (4) | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 (5) | 0
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0
Ulceration (General disorders) | 0 | 0 | 1 (1) | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 1 (2) | 0
Vaginal mucositis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 (2)
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Vision - blurred vision (Eye disorders) | 0 | 0 | 3 (7) | 0
Vision - flashing lights/floaters (Eye disorders) | 0 | 0 | 0 | 1 (1)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 5 (8) | 3 (3) | 8 (22) | 2 (3)
Watery eye (Eye disorders) | 0 | 0 | 1 (1) | 0
Weight gain (Investigations) | 0 | 0 | 1 (5) | 0
Weight loss (Investigations) | 0 | 3 (3) | 8 (10) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No